CLINICAL TRIAL: NCT04917640
Title: Accelerated Partial Breast Irradiation (PBI) With Stereotactic Body Radiation Therapy (SBRT) or Intensity Modulated Radiation Therapy (IMRT)
Brief Title: Registry for Accelerated Partial Breast Irradiation With (SBRT) or (IMRT)
Status: Withdrawn | Type: Observational
Why Stopped: A revised study has been listed here for us.
Sponsor: GenesisCare USA (Other)
Responsible Party: Sponsor
Other Study IDs: APBI Registry
Record Dates: First submitted 2021-05-24; First posted 2021-06-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SBRT: Patients treated with Stereotactic Body Radiation Therapy (SBRT)
  Interventions: Radiation: Radiation Therapy
- IMRT: Patients treated with Intensity Modulated Radiation Therapy (IMRT)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Either SBRT or IMRT radiation therapy

SUMMARY:
This is a registry study that will be used to evaluate external beam radiation therapy methods for the accelerated treatment of breast cancer. Patients are being asked to take part in this registry because they have breast cancer and desire treatment with accelerated partial breast irradiation to be delivered by external beam methods.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 50 years old Low to intermediate DCIS Tumor size < or = to 2cm

Exclusion Criteria:

* BRCA positive Lobular histology Angiolymphatic invasion

Ages: 50 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women 50 years old or older who have been diagnosed with low to intermediate DCIS
Study Population: Women with greater than or equal to 50 years old and who have been diagnosed with Low to intermediate DCIS
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment and toxicity-related adverse events as assessed by CTCAE v4.0". | Through study completion, an average of 12 months
  Toxicity will be assessed using the CTCAEv4.0 and recorded.

SECONDARY OUTCOMES:
Number of participants with ipsilateral breast recurrence | Through study completion, an average of 12 months
  Number of participants with pathologically confirmed ipsilateral breast recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Salenius, MPH, Study Director — Fundacion GenesisCare
Locations (1):
- GenesisCare USA, Stuart, Florida, United States

IPD SHARING:
Plan to Share IPD: No